CLINICAL TRIAL: NCT02580474
Title: The Safety and Efficacy of Daclatasvir and Asunaprevir With Chronic HCV Genotype 1b Infection and Chronic Renal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Myeong Jun Song (Other)
Collaborators: Bristol-Myers Squibb (Industry); Soonchunhyang University Hospital (Other); Dankook University (Other); Chungnam National University Hospital (Other); Konyang University Hospital (Other); Eulji University Hospital (Other); Saint Vincent's Hospital, Korea (Other); Konkuk University Hospital (Other); Cheongju St. Mary's Hospital, Cheongju, Korea (Other); Severance Hospital (Other); Korea University Guro Hospital (Other); Eulji General Hospital (Other)
Responsible Party: Sponsor-Investigator, Myeong Jun Song, Assistant Professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI447-118
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daclatasvir plus Asunaprevir (Experimental)
  Interventions: Drug: Daclatasvir plus Asunaprevir

INTERVENTIONS:
Drug: Daclatasvir plus Asunaprevir

SUMMARY:
Safety and Efficacy of DAAs (Daclatasvir+Asunaprevir) in patients with chronic hepatitis C and chronic renal failure will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA Positive and Genotype 1b
* No history or signs or symptoms of decompensated liver disease or hepatocellular carcinoma within 6 months
* A patient who is on dialysis, or if not MDRD eGFR<30ml/min
* HCV treatment history: HCV treatment-naive participants, defined as never having received HCV treatment with any approved or investigational drug (including vaccines); OR HCV treatment-experienced, defined as having received previous HCV treatment with any (pegylated) interferon ([Peg]IFN)-based drug regimen (with or without ribavirin [RBV] and not including a direct-acting antiviral agent [DAA]). Last dose in this previous HCV treatment course should have occurred at least 2 months prior to screening
* No baseline mutation NS5A polymorphism including L31F/I/M/V and Y93H

Exclusion Criteria:

* A patient who having received Daclatasvir or Asunaprevir
* Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study
* Evidence of a medical condition contributing to chronic liver disease other than HCV or seropositive for HIV
* Diagnosed or suspected hepatocellular carcinoma or other malignancies
* Any history of, or current evidence of, clinical hepatic decompensation (e.g., ascites, encephalopathy or variceal hemorrhage)
* Received solid organ or bone marrow transplant
* Current alcohol or substance abuse judged by the investigator to potentially interfere with subject compliance
* Significant renal, cardiovascular, pulmonary, or neurological disease and uncontrolled diabetes or hypertension in the opinion of the investigator
* Known hypersensitivity to study drugs, metabolites, or formulation excipients
* Who has taken investigational drugs within 2 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
the proportion of subjects with plasma HCV RNA levels below 15 IU/mL at Week 12 After End of Treatment | 36 Week

SECONDARY OUTCOMES:
To evaluate the percentage of subjects with Sustained Virologic Response at Week 12 After End of Treatment | 36 Week
Percentage of subjects with ALT normalization at each visit from the baseline | 4, 12, 24, 36 week
Change in HCV RNA at each visit from the baseline | 4, 12, 24, 36 week
Percentage of subjects who experience viral breakthrough at each visit from the baseline | 4, 12, 24, 36 week
Percentage of subjects who shows Tolerability of Daclatasvir and Asunaprevir at each visit from | 4, 12, 24, 36 week

CONTACTS AND LOCATIONS:
Locations (1):
- Myeong Jun Song, Daejeon, South Korea

REFERENCES:
- [Derived] Lee BS, Song MJ, Kwon JH, Lee TH, Jang JW, Kim SH, Lee SH, Kim HS, Kim JH, Kim SB, Ko SY, Song DS. Efficacy and Safety of Daclatasvir and Asunaprevir in Patients with Hepatitis C Virus Genotype 1b Infection on Hemodialysis. Gut Liver. 2019 Mar 15;13(2):191-196. doi: 10.5009/gnl18240. PMID 30400729